CLINICAL TRIAL: NCT00860327
Title: Excitation-contraction Coupling in Human Ventricle Development
Brief Title: Examining Developmental Changes in Heart Contractions of Children With Congenital Heart Defects
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary Wagner, Assistant Professor, Emory University
Other Study IDs: IRB00007244; R01HL088488 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Hypoplastic Left Heart Syndrome; Tetralogy of Fallot
Keywords: Pediatric Heart Disease; Congenital Heart Disease; Congenital Heart Defects; Developmental Biology; Contractile Function
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Tetralogy of Fallot; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ventricular tissue, that would have been discarded, and was removed during surgery as part of the necessary repair for congenital heart defects
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Newborns: Newborns with hypoplastic left heart syndrome who are receiving a right ventricle to pulmonary artery shunt as first stage palliation.
- Infants: Infants who are undergoing complete repair for tetralogy of Fallot or similar pathology.

SUMMARY:
Children who are born with heart defects undergo surgery when they are infants to correct the defects. However, many treatments that are used in pediatric heart patients were originally developed for adults and may not be the best option for children. This study will analyze tissue samples from newborns and infants undergoing surgery for heart defects to learn more about how a child's heart develops during the first year of life. This information may help to identify possible treatments geared specifically for the pediatric heart patient.

DETAILED DESCRIPTION:
Congenital heart defects are abnormalities or problems with the structure of the heart that are present at birth. Examples of congenital heart defects include hypoplastic left heart syndrome, which is a condition that occurs when the left side of the heart does not develop completely, and tetralogy of Fallot, which is a condition that involves four specific types of structural defects within the heart. Many advances have been made in recent years in the field of pediatric heart surgery, and children who are born with congenital heart defects are now able to undergo heart surgery as infants to repair the defects. However, very little is known about the differences between how an infant's heart functions and how an adult's heart functions. Thus, most of the therapies that are used to treat children with heart defects were originally developed for adults and may not be the best option for infants and young children. The purpose of this study is to gain a better understanding of how the heart changes during a child's first year of life, from being a newborn less than 1 week old to being an infant 3 to 12 months old.

During surgical repair of congenital heart defects, tissue from the ventricular structures of the heart is sometimes removed as part of the surgery. In this study, researchers will examine ventricular tissue removed during the surgical procedures of newborns with hypoplastic left heart syndrome and infants with tetralogy of Fallot. Study researchers will compare the newborn and infant tissue samples in terms of their differences in excitation-contraction coupling, also referred to as contraction response. Excitation-contraction coupling in the heart is the process wherein electrical activity of the heart is translated into contraction of the heart muscle, which then results in pumping of the blood out to the body. Study researchers will also examine how calcium, which is required for heart contraction, flows in and out of heart cells to determine whether the process differs among newborns and infants. Acquiring data on both excitation-contraction coupling and the role of calcium is important because increasing the strength of heart contractions is a key component of treatment options for children with congenital heart defects.

This study has been granted a waiver of consent as de-identified tissue will be collected from waste samples. The number of participants represents the number of samples collected.

ELIGIBILITY:
Inclusion Criteria:

* Newborns less than 1 week of age with hypoplastic left heart syndrome
* Infants between 3 to 12 months of age with tetralogy of Fallot
* Requires removal of ventricular tissue during surgery as part of the repair for a congenital heart defect

Exclusion Criteria

- Children > 12 months of age

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing surgery for repair of congenital heart defects.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2007-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Calcium handling assay | At time of aquisition
  Calcium handling will be assayed in tissue or cells by patch clamp, imaging or protein level measurement and will be done at the time the tissue is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Mary B. Wagner, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Department of Pediatrics, Atlanta, Georgia, United States

REFERENCES:
- [Result] Wiegerinck RF, Cojoc A, Zeidenweber CM, Ding G, Shen M, Joyner RW, Fernandez JD, Kanter KR, Kirshbom PM, Kogon BE, Wagner MB. Force frequency relationship of the human ventricle increases during early postnatal development. Pediatr Res. 2009 Apr;65(4):414-9. doi: 10.1203/PDR.0b013e318199093c. PMID 19127223